CLINICAL TRIAL: NCT01685346
Title: Biofeedback Training in Patients With Advanced Lung Cancer - A Pilot Study
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Research Cancelled
Sponsor: Case Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: CASE6512; 12-874 (Other: Cleveland Clinic IRB)
Record Dates: First submitted 2012-09-10; First posted 2012-09-14 (Estimated); Last update posted 2015-07-10 (Estimated); Status verified 2015-07

CONDITIONS: Advanced (Stage IV) Non-small Cell Lung Cancer (NSCLC)
Keywords: advanced (stage IV) non-small cell lung cancer (NSCLC); biofeedback-mediated stress management (BFSM)
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Biofeedback (Experimental): biofeedback-mediated stress management (BFSM)
  Interventions: Behavioral: biofeedback-mediated stress management (BFSM)

INTERVENTIONS:
Behavioral: biofeedback-mediated stress management (BFSM) — Therapist and study assistant meet with patient, attach sensors, record physiologic variables and train the patient in relaxation techniques including deep breathing, guided imagery, progressive muscle relaxation, autogenics. Patient is given a handheld thermometer to take home and practice self-regulation between visits, along with a recording sheet to indicate how often practice occurs.

SUMMARY:
This is a pilot study to test the hypothesis that biofeedback-mediated stress management (BFSM) training can be used to reduce distress and enhance quality of life in patients with non-small cell lung cancer (NSCLC). Most patients with advanced NSCLC have significant physical symptoms, but even those who do not have physical symptoms have high levels of anxiety and depression.

DETAILED DESCRIPTION:
Biofeedback-mediated stress management (BFSM) involves helping patients to visualize the reactions which their own bodies have to stressful situations (increased heart rate, increased skin conductance, increased muscle tension, decreased digital peripheral temperature, decreased heart rate variability) and then teaching them to control these reactions, using standard stress management and relaxation techniques, coupled with computerized physiological feedback. The feedback helps patients to understand that deep relaxation is helping their bodies as well as their minds. Several small studies of BFSM training in cancer populations have been successful at helping with side effects of chemotherapy and radiation, but the effects of BFSM on distress and quality of life (QOL), particularly in NSCLC patients, have not been studied.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a new diagnosis of advanced (stage IV) non-small cell lung cancer (NSCLC)
* ECOG performance status 0-1.
* Plan to receive care at the Taussig Cancer Center.

Exclusion Criteria:

* Non-local patients, who will not have the ability to return for 8 study visits.
* Patients who are unable to speak and understand English readily,
* Patients with significant cognitive impairment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2012-10; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Number of patients that are able to return for eight visits of BFSM | 16 weeks
  Keep track of how many visits the patients attend, how many they cancel, and what other difficulties are encounter in getting them to return for eight visits.

SECONDARY OUTCOMES:
Number of patients able to complete the Quality of Life (QOL) questionnaires | 16 weeks
Assess changes in distress thermometer from baseline | 16 weeks
  Distress Thermometer questionnaire using a scale of 0-10. O meaning no distress and 10 meaning extreme distress.
Change from baseline on the FACT-lung questionnaire | 16 weeks
  Physical, social/family, emotional, and functional well-being on a 0-4 scale. O being not at all and 4 being very much.
Change from baseline of the Hospital Anxiety and Depression Scale (HADS) | 16 weeks
  Questionnaire to determine the levels of anxiety and depression that a patient is experiencing. The HADS is a fourteen item scale that generates ordinal data.
Change from baseline of the Patient Health Questionnaire (PHQ-*8) | 16 weeks
  8-Item depression health questionnaire based on a scale from 0-3. 0 meaning not at all and 3 meaning nearly every day.
Change in baseline of digital peripheral temperature | 16 weeks
  Compare the baseline measurement during the first five minutes of the session, the peak response to mental stress during the next ten minutes of the session, and the response during the self-relaxation period following the mental stress. An improvement would indicate success with biofeedback.
Change in baseline of skin conductance | 16 weeks
  Compare the baseline measurement during the first five minutes of the session, the peak response to mental stress during the next ten minutes of the session, and the response during the self-relaxation period following the mental stress. An improvement would indicate success with biofeedback.
Change from baseline of Electromyography (EMG) | 16 weeks
  Compare the baseline measurement during the first five minutes of the session, the peak response to mental stress during the next ten minutes of the session, and the response during the self-relaxation period following the mental stress. An improvement would indicate success with biofeedback.
Change from baseline of respiratory rates | 16 weeks
  Compare the baseline measurement during the first five minutes of the session, the peak response to mental stress during the next ten minutes of the session, and the response during the self-relaxation period following the mental stress. An improvement would indicate success with biofeedback.
Change from baseline of heart rates | 16 weeks
  Compare the baseline measurement during the first five minutes of the session, the peak response to mental stress during the next ten minutes of the session, and the response during the self-relaxation period following the mental stress. An improvement would indicate success with biofeedback.

CONTACTS AND LOCATIONS:
Overall Officials: Nathan Pennell, MD, Principal Investigator — Cleveland Clinic Taussig Cancer Center, Case Comprehensive Cancer Center
Locations (1):
- Cleveland Clinic Taussig Cancer Center, Case Comprehensive Cancer Center, Cleveland, Ohio, United States